CLINICAL TRIAL: NCT04231630
Title: A Single Patient Observational Trial of an Exclusive Human Milk Diet to Provide and Evaluate Growth in a Single Infant at Home With Complex Congenital Heart Disease
Brief Title: Outpatient Exclusive Human Milk Diet for Single Infant With Complex Congenital Heart Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Texas at Austin (Other)
Collaborators: Prolacta Bioscience (Industry)
Responsible Party: Principal Investigator, Steven Abrams, Professor, University of Texas at Austin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-11-0001
Record Dates: First submitted 2020-01-09; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Growth Delay

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Observational Case (Other): 1 infant will be enrolled as an observational case. Will receive an exclusive human milk diet at home.
  Interventions: Other: Prolacta

INTERVENTIONS:
Other: Prolacta — Will receive outpatient supplementation with donor human milk product added to mother's own milk

SUMMARY:
A single patient observational trial to evaluate growth velocity and clinical outcomes of an infant status post cardiac surgery who has failed to grow well and demonstrated intolerance to cow milk-based and elemental formulas and fortifiers on a 100% human milk diet including a human milk based human milk fortifier formulated for term infants fluid restricted due to surgically correctable congenital conditions.

DETAILED DESCRIPTION:
A single patient observational study to evaluate growth velocity and clinical outcomes of an infant status post cardiac surgery who has failed to grow well and demonstrated intolerance to cow milk-based and elemental formulas and fortifiers on a 100% human milk diet. Human milk is defined as expressed human milk or donor milk and its derivatives, human milk-based fortifier and human milk caloric fortifier.

The study hypothesis is that this infant if fed an exclusive human milk diet will have improved growth in part due to data greater tolerability of the diet.

It is estimated that the study will require 90 days to complete. Growth in safety observations will be collected only during the time the patient is receiving the diet.

The primary objective is to evaluate growth velocity (weight velocity [g/kg/day] of a single infant receiving a 100% human milk diet including a human milk based human milk fortifier formulated for term infants who are fluid restricted due to surgically correctable congenital conditions. This will be compared to the infant's growth velocity prior to the initiation of said diet.

ELIGIBILITY:
Inclusion Criteria:

* Complex congenital heart disease in presence of poor linear and head circumference growth and unable to tolerate cow's milk protein

Exclusion Criteria:

* n/a

Ages: 6 Months to 1 Year | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-05-30 (Estimated)

PRIMARY OUTCOMES:
Growth | through study completion, approximately 6 months
  Weight velocity

SECONDARY OUTCOMES:
Linear growth | through study completion, approximately 6 months
  Length gain
Head circumference growth | through study completion, approximately 6 months
  Head circumference growth

CONTACTS AND LOCATIONS:
Locations (1):
- Dell Medical School, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No